CLINICAL TRIAL: NCT00768807
Title: Structural and Functional Left Ventricular Remodelling in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Wercules Antonio Alves de Oliveira, Dr., Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ECOera-03
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham CPAP (Sham Comparator): Patients submitted to SHAM CPAP use for 06 months
  Interventions: Device: CPAP (continuous positive airway pressure)
- CPAP (Active Comparator): OSA patients submitted to 06 months of CPAP treatment
  Interventions: Device: CPAP (continuous positive airway pressure)

INTERVENTIONS:
Device: CPAP (continuous positive airway pressure) — Patients treated by CPAP for 06 months

SUMMARY:
The purpose of this study is to determine whether patients with obstructive sleep apnea have any changes in left ventricular function and structure after 06 months of continuous positive airway pressure treatment.

DETAILED DESCRIPTION:
Several studies have been suggesting that Obstructive Sleep Apnea contributes to deterioration of left ventricular diastolic function. It may be associated to increased risk of cardiovascular events. We hypothesized that morphological and functional left ventricular changes might be reverted after treatment with Continuous positive airway pressure.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-hypopnea index higher than 5 events per hour

Exclusion Criteria:

* Body mass index higher than 40 kg/m2

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Improvement of left ventricular diastolic echo variable | 06 months

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Sono/AFIP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Oliveira W, Campos O, Cintra F, Matos L, Vieira ML, Rollim B, Fujita L, Tufik S, Poyares D. Impact of continuous positive airway pressure treatment on left atrial volume and function in patients with obstructive sleep apnoea assessed by real-time three-dimensional echocardiography. Heart. 2009 Nov;95(22):1872-8. doi: 10.1136/hrt.2009.173625. Epub 2009 Jul 29. PMID 19643769